CLINICAL TRIAL: NCT04979546
Title: Using Patient-Reported Outcomes To Improve the Care of People With Multiple Sclerosis: A Randomized Trial
Brief Title: Using Patient-Reported Outcomes To Improve the Care of People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00111593
Record Dates: First submitted 2021-07-06; First posted 2021-07-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Anxiety; Depression; Patient Satisfaction
Keywords: patient reported outcome measures, consultant satisfaction shared decision-making
MeSH Terms: conditions — Multiple Sclerosis; Anxiety Disorders; Depression; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Intervention group: All participants randomized to the intervention group will be asked to complete PROM questionnaires at baseline, 6 months and 12 months (12 month study duration). Their treating neurologist will view the participant scores in addition to the text response to the 3-item prompt.
  Control group: those in the control group will complete the same questionnaires at baseline and at 12 months. Additionally, the treating neurologist will only be prompted to view the text response to the 3-item prompt, and will not be able to access the PROM questionnaire scores for participants in the control group.
Who Masked: Outcomes Assessor
Masking Description: The participants will know if they have been randomized to the intensive arm or the control arm, by whether they are completing PROMs every 6 months versus 1 year. The treating neurologists will know which arm their patients are enrolled into by whether they receive all PROM measurements every 6 months on their patients versus solely a text response of the "top 3 things their patient would like their neurologist to know" at that time.
  Data analysis will be anonymized and aggregated for the research team in analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive PROMs Intervention Arm (Experimental): The intervention group will be asked to complete PROM questionnaires at baseline, 6 months, and 12 months via an online web-based delivery system. The treating neurologist will be prompted to view the text response to the 3-item prompt in addition to the PROM questionnaire scores for participants in the interventional group. Treating neurologist will also be alerted if participates reach certain critical threshold scores or decrement on their PROM questionnaires. Participants randomized to the intervention group will be asked to complete CSQ and CollaboRATE questionnaires at baseline and at 12 months.
  Interventions: Other: Intensive Use of Patient Reported Outcome Measures and Open PROM Availability to Treating Neurologist
- Control Arm (Active Comparator): The control group will be asked to complete PROM questionnaires at baseline and 12 months via an online web-based delivery system. The treating neurologist will only be prompted to view the text response to the 3-item prompt, and will not be able to access the PROM questionnaire scores for participants in the control group (unless critical values are reached on questionnaires - see below). Treating neurologist will also be alerted if participates reach certain critical threshold scores or decrement on their PROM questionnaires. Participants randomized to the intervention group will be asked to complete CSQ and CollaboRATE questionnaires at baseline and at 12 months.
  Interventions: Other: Conservative Use of Patient Reported Outcome Measures and Blinded PROM Availability to Treating Neurologist

INTERVENTIONS:
Other: Intensive Use of Patient Reported Outcome Measures and Open PROM Availability to Treating Neurologist — Baseline, 6 months, and 12 months administration of HADS, EQ5D, MFIS, PDDS, PHQ-9 questionnaires in addition to Open ended text response to (limit 280 characters) "What are the top 3 things you would like your MS Neurologist to know about you right now?"
  Additionally, the treating neurologist will be prompted to view the text response to the 3-item prompt in addition to the PROM questionnaire scores for participants in the interventional group.
  Arms: Intensive PROMs Intervention Arm
Other: Conservative Use of Patient Reported Outcome Measures and Blinded PROM Availability to Treating Neurologist — Baseline and 12 months administration of HADS, EQ5D, MFIS, PDDS, PHQ-9 questionnaires in addition to Open ended text response to (limit 280 characters) "What are the top 3 things you would like your MS Neurologist to know about you right now?"
  Additionally, the treating neurologist will only be prompted to view the text response to the 3-item prompt, and will not be able to access the PROM questionnaire scores for participants in the control group.
  Arms: Control Arm

SUMMARY:
The proposed trial is a prospective, randomized (1:1) trial plan examining whether more routine and frequent measurement of Patient Related Outcome Measures (PROMs) in the care of patients with MS improves patient depression and anxiety outcomes in addition to patient care satisfaction. The investigators plan to randomize people with MS (PwMS) to an intensive arm of filling out patient reported outcome measures every 6 months, with communication to their neurologist about their scores, versus a control arm, where participants fill out patient reported outcomes less frequently (annually) and their scores are not released to their MS Clinic/Neurologist. The primary outcome is to see if more frequent PROM completion leads to less depression and anxiety for people with MS. The investigators also plan to measure their satisfaction of care with their MS Clinic/neurologist and satisfaction in a shared decision-making process.

Whether this improves care in patients with MS is currently unknown, and the investigators want to explore this with the current study. The investigators plan to randomize people with MS (PwMS) to an intensive arm of filling out patient reported outcome measures every 6 months, with communication to their neurologist about their scores, versus a control arm, where participants fill out patient reported outcomes less frequently (annually) and their scores are not released to their MS Clinic/Neurologist. The primary outcome is to see if more frequent PROM completion leads to less anxiety for people with MS. The investigators also plan to measure their satisfaction of care with their MS Clinic/neurologist and satisfaction in a shared decision-making process.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a disease that can affect physical, cognitive, psychological, and social functioning. Patient reported outcomes measures (PROMs) are playing an increasingly important role in healthcare as they give patients the opportunity to describe the quality and the impact of care from their perspective in a consistent and systematic way. PROMs are important in optimizing the management of people with MS (PwMS) in providing the patient's perspective of their disease. Additionally, use of PROMs between clinic visits could provide real-time information about how well patients are doing between visits, in a disease with episodic disability and with symptoms that fluctuate over time. Electronic data capture could help overcome these difficulties, as patients will have the flexibility to provide the information from anywhere and the data will automatically be saved in an electronic database that can be accessed anytime by patients and their healthcare providers. This will allow patients to be fully informed about their condition, be more engaged in their care, track their progress, and receive any notifications or alerts regarding their care. It will also allow healthcare providers to systematically track the patient's progress, better prepare for their visit and provide care based on their individual needs - the epitome of patient-centred care. Even though such information could help clinicians provide patient-centred care and patients track their progress, it is not collected on a routine basis during clinical care due to time limitations, and system issues within clinics amongst other factors.

The investigators' objective is to evaluate the impact of the systematic and more frequent use of PROMs in PwMS on depression and anxiety levels and satisfaction with care.

The investigators will be conducting a randomized controlled trial with the participant as the unit of randomization. They will include PwMS (relapsing-remitting, secondary progressive, primary progressive, etc.) who are being managed by an Alberta-based neurologist in the Northern and Central regions. Recruited participants will be randomized 1:1 to an interventional group or a control group. The interventional group will complete PROM questionnaires at baseline, 6 months, and 12 months in addition to their treating neurologist alerted to and having access to their questionnaire results and text response to the question "What are the top 3 things you would like your MS Neurologist to know about you right now?"; the control group will complete PROM questionnaires at baseline and at 12 months, and while their neurologist will be able to view their text response to the question "What are the top 3 things you would like your MS Neurologist to know about you right now?", the neurologist will not have routine access to their PROM questionnaire results.

All participants will be asked to complete the following validated PROMs questionnaires at intervals designated by their assigned experimental group:

1. Hospital Anxiety and Depression Scale (HADS) score
2. Quality of Life as measured by EuroQol Five-Dimensions (EQ5D) questionnaire
3. Fatigue as measured by Modified Fatigue Impact Scale (MFIS)
4. The Patient Determined Disease Steps (PDDS)
5. Patient Health Questionnaire-9 (PHQ-9)
6. Open ended text response to (limit 280 characters) "What are the top 3 things you would like your MS Neurologist to know about you right now?"

For both groups, critical absolute scores or decrement in subsequent scores as measured by the aforementioned questionnaires will trigger an automated secured email alert to the patient's treating neurologist. Critical PROM scores are defined as:

1. EQ5D index value ≤ 0.48 at any time OR decrease in index value ≥ 0.26 on subsequent testing to capture those with a substantial decrease in their score over time.
2. MFIS absolute total score ≥ 58 at any time OR increase in absolute total score ≥ 17 on subsequent testing to capture those with a substantial increase in their score over time.
3. HADS score with an absolute score ≥ 11 in either depression or anxiety category at any time, OR increase in depression or anxiety score ≥ 4 on subsequent testing.
4. PDDS ≥ 3 at first testing - trigger to notify with gait impairment but not requiring aid yet, OR increase of score ≥ 1 on subsequent measurements.
5. PHQ-9 score of ≥ 10 at any time OR increase in score by ≥ 6 on subsequent testing.

All groups will also be asked to complete the Consultation Satisfaction Questionnaire (CSQ) as a measure of provider satisfaction, and the CollaboRATE survey as a measure of shared decision-making, at baseline, and at end of the study at 12 months.

Patient providers will additionally be asked to fill out an exit survey at the end of the study, assessing their opinion on the subjective effectiveness of implementing PROM questionnaires and the open ended text response to care of PwMS. Seven questions assessed on a Likert scale from 1-5 (strongly disagree to strongly agree), one question as a multiple choice response, and one open ended response will be assessed on the exit survey.

ELIGIBILITY:
Inclusion Criteria:

* Persons with multiple sclerosis [relapsing-remitting, secondary progressive, primary progressive, etc.] being managed by a Northern or Central Alberta-based neurologist.
* Able/willing to complete informed consent and the questionnaires.
* Able to use a computer.
* Greater or equal to the age of 18 years old.
* English-speaking.

Exclusion Criteria:

* Unwilling/unable to provide consent.
* Unwilling/unable to complete the questionnaires.
* Does not speak English.
* Under the age of 18.
* Has a central nervous system inflammatory disorder other than MS.
* PwMS not being managed by the participating neurologist (a neurologist practicing in Northern and Central Alberta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Difference in Change in Depression score in the Hospital Anxiety and Depression Scale (HADS-D) scores | 12 months
  Hospital Anxiety & Depression Scale (D subcategory for depression levels, A subcategory for anxiety levels). This is a common depression and anxiety measurement instrument used in multiple sclerosis (Jones et al, PLoS One 2012). Minimum score is 0, and maximum score is 21. Higher scores indicate worse outcome.
  Three papers report total HADS scores in PwMS. Using the information from Honarmand and Feinstein (Mult Scler, 2009) [Baseline scores and standard deviation (SD)] and the following assumptions 90% power and a two-sided alpha of 0.05, a total sample size of 200 (100 in each group) was required to detect 1.5 difference between the intervention and the control groups. This sample size was inflated to 220 to account for possible dropouts, losses to follow-up and withdrawals of consent.
Difference in Change in Anxiety score in the Hospital Anxiety and Depression Scale (HADS-A) scores | 12 months
  Hospital Anxiety & Depression Scale (D subcategory for depression levels, A subcategory for anxiety levels). This is a common depression and anxiety measurement instrument used in multiple sclerosis (Jones et al, PLoS One 2012). Minimum score is 0, and maximum score is 21. Higher scores indicate worse outcome.
  Three papers report total HADS scores in PwMS. Using the information from Honarmand and Feinstein (Mult Scler, 2009) [Baseline scores and standard deviation (SD)] and the following assumptions 90% power and a two-sided alpha of 0.05, a total sample size of 200 (100 in each group) was required to detect 1.5 difference between the intervention and the control groups. This sample size was inflated to 220 to account for possible dropouts, losses to follow-up and withdrawals of consent.

SECONDARY OUTCOMES:
Difference in Change in the Euro Quality of Life Measurement (EQ5D) | 12 months
  The EQ5D quality of life measure is used in the MS population (Kuspinar & Mayo, Pharmacoeconomics 2014), and is the main quality of life measure preferred by Alberta Health Services. There is a descriptive element to the EQ5D that represents values around the level of reported problems in each of the 5 domains, with higher scores being worse. The 5 domains are around (1) mobility; (2) self-care; (3) usual activities; (4) pain/discomfort; and (5) anxiety/depression. The index is calculated by deducting the appropriate weights from 1 and comparing to population norms in a value set.
Difference in Change in the Modified Fatigue Impact Scale (MFIS) score | 12 months
  Fatigue is one of the most common symptoms for people with MS. The MSIF is a standard, validated measurement of fatigue in MS (Fisk et al, Can J Neurol Sci 1994). The MFIS is a self-report instrument in which participants are asked to rate how often fatigue has affected them in the previous 4 weeks in relation to statements (0 = never to 4 = almost always). Items on the MFIS can be aggregated into subscales (physical, cognitive and psychosocial) as well as into a total MFIS score. The total MFIS score can be a minimum of 0 to 84, computed by adding the scores on the physical, cognitive and psychosocial subscales.
Scores on Qualitative Consultant Satisfaction Questionnaire (CSQ) | 12 months
  Participants' satisfaction with the level of care provided to them will be measured at 6 months using the validated Consultant Satisfaction Questionnaire (CSQ) (Baker, Br J Gen Pract 1990). CSQ consists of 18 Likert scale questions, ranging from 1= strongly disagree to 5 = strongly agree, with the higher score indicating higher patient satisfaction. Satisfaction with healthcare provider care will be measured by the overall mean score of the consultation satisfaction questionnaire (CSQ) completed at the 6 month follow-up visit. The CSQ is a self-administered tool with 18 questions using a 5-point Likert scale, ranging from strongly agree to strongly disagree. It measures 3 factors of the healthcare provider interaction: (1) professional aspects; (2) depth of patient relationship with provider; and (3) perceived length of consultation. Higher scores indicate higher satisfaction.
The Patient Determined Disease Steps (PDDS) Stability of Score | 12 months
  The Patient Determined Disease Steps (PDDS) score is a patient reported measure of disability in multiple sclerosis, that has been validated in comparing to the gold standard of MS disability measurement, the Expanded Disability Status Score (EDSS). (Learmouth et al, BMC Neurology 2013; Hohol et al, Mult Scler. 1999)
Difference in Change in the Patient Health Questionnaire-9 (PHQ-9) | 12 months
  PwMS have a high prevalence of depression. The Patient Health Questionnaire-9 (PHQ-9) is a frequently used measure of depression in the MS population. It has been shown to be valid in the MS population (Sjonnesen et al, Postgraduate Medicine 2015)
Difference in change in the CollaboRATE shared decision-making survey | 12 months
  The CollaboRATE is a brief, patient survey that focuses on the patient's perceived input and satisfaction with the shared decision-making process around their health decisions with their health care providers. (Elwyn et al, Patient Educ Couns 2013; Forcino et al, Health Expectations 2018)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers. We plan to analyze outcomes and publish the data as aggregated, anonymized data.

REFERENCES:
- [Background] Baker R. Development of a questionnaire to assess patients' satisfaction with consultations in general practice. Br J Gen Pract. 1990 Dec;40(341):487-90. PMID 2282225
- [Background] Fiest KM, Walker JR, Bernstein CN, Graff LA, Zarychanski R, Abou-Setta AM, Patten SB, Sareen J, Bolton JM, Marriott JJ, Fisk JD, Singer A, Marrie RA; CIHR Team Defining the Burden and Managing the Effects of Psychiatric Comorbidity in Chronic Immunoinflammatory Disease. Systematic review and meta-analysis of interventions for depression and anxiety in persons with multiple sclerosis. Mult Scler Relat Disord. 2016 Jan;5:12-26. doi: 10.1016/j.msard.2015.10.004. Epub 2015 Oct 19. PMID 26856938
- [Background] Fisk JD, Pontefract A, Ritvo PG, Archibald CJ, Murray TJ. The impact of fatigue on patients with multiple sclerosis. Can J Neurol Sci. 1994 Feb;21(1):9-14. PMID 8180914
- [Background] Forbes A, While A, Mathes L, Griffiths P. Health problems and health-related quality of life in people with multiple sclerosis. Clin Rehabil. 2006 Jan;20(1):67-78. doi: 10.1191/0269215506cr880oa. PMID 16502752
- [Background] Honarmand K, Feinstein A. Validation of the Hospital Anxiety and Depression Scale for use with multiple sclerosis patients. Mult Scler. 2009 Dec;15(12):1518-24. doi: 10.1177/1352458509347150. Epub 2009 Nov 13. PMID 19965520
- [Background] Jones KH, Ford DV, Jones PA, John A, Middleton RM, Lockhart-Jones H, Osborne LA, Noble JG. A large-scale study of anxiety and depression in people with Multiple Sclerosis: a survey via the web portal of the UK MS Register. PLoS One. 2012;7(7):e41910. doi: 10.1371/journal.pone.0041910. Epub 2012 Jul 30. PMID 22860028
- [Background] Kuspinar A, Mayo NE. A review of the psychometric properties of generic utility measures in multiple sclerosis. Pharmacoeconomics. 2014 Aug;32(8):759-73. doi: 10.1007/s40273-014-0167-5. PMID 24846760
- [Background] Montanari E, Rottoli M, Maimone D, Confalonieri P, Plewnia K, Frigo M, Francia A, Pala A, Losignore NA, Ragonese P, Veneziano A; POSIDONIA study group. A 12-month prospective, observational study evaluating the impact of disease-modifying treatment on emotional burden in recently-diagnosed multiple sclerosis patients: The POSIDONIA study. J Neurol Sci. 2016 May 15;364:105-9. doi: 10.1016/j.jns.2016.02.047. Epub 2016 Feb 20. PMID 27084226
- [Background] Nourbakhsh B, Julian L, Waubant E. Fatigue and depression predict quality of life in patients with early multiple sclerosis: a longitudinal study. Eur J Neurol. 2016 Sep;23(9):1482-6. doi: 10.1111/ene.13102. Epub 2016 Jul 14. PMID 27416110
- [Background] Ponzio M, Tacchino A, Vaccaro C, Traversa S, Brichetto G, Battaglia MA, Uccelli MM. Unmet needs influence health-related quality of life in people with multiple sclerosis. Mult Scler Relat Disord. 2020 Feb;38:101877. doi: 10.1016/j.msard.2019.101877. Epub 2019 Nov 29. PMID 31812039
- [Background] Puhan MA, Frey M, Buchi S, Schunemann HJ. The minimal important difference of the hospital anxiety and depression scale in patients with chronic obstructive pulmonary disease. Health Qual Life Outcomes. 2008 Jul 2;6:46. doi: 10.1186/1477-7525-6-46. PMID 18597689
- [Background] Puhan MA, Gaspoz JM, Bridevaux PO, Schindler C, Ackermann-Liebrich U, Rochat T, Gerbase MW. Comparing a disease-specific and a generic health-related quality of life instrument in subjects with asthma from the general population. Health Qual Life Outcomes. 2008 Feb 15;6:15. doi: 10.1186/1477-7525-6-15. PMID 18279510
- [Background] Amankwah N, Marrie RA, Bancej C, Garner R, Manuel DG, Wall R, Fines P, Bernier J, Tu K, Reimer K. Multiple sclerosis in Canada 2011 to 2031: results of a microsimulation modelling study of epidemiological and economic impacts. Health Promot Chronic Dis Prev Can. 2017 Feb;37(2):37-48. doi: 10.24095/hpcdp.37.2.02. PMID 28273039
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Hobart J, Bowen A, Pepper G, Crofts H, Eberhard L, Berger T, Boyko A, Boz C, Butzkueven H, Celius EG, Drulovic J, Flores J, Horakova D, Lebrun-Frenay C, Marrie RA, Overell J, Piehl F, Rasmussen PV, Sa MJ, Sirbu CA, Skromne E, Torkildsen O, van Pesch V, Vollmer T, Zakaria M, Ziemssen T, Giovannoni G. International consensus on quality standards for brain health-focused care in multiple sclerosis. Mult Scler. 2019 Nov;25(13):1809-1818. doi: 10.1177/1352458518809326. Epub 2018 Nov 1. PMID 30381987
- [Background] Forcino RC, Barr PJ, O'Malley AJ, Arend R, Castaldo MG, Ozanne EM, Percac-Lima S, Stults CD, Tai-Seale M, Thompson R, Elwyn G. Using CollaboRATE, a brief patient-reported measure of shared decision making: Results from three clinical settings in the United States. Health Expect. 2018 Feb;21(1):82-89. doi: 10.1111/hex.12588. Epub 2017 Jul 5. PMID 28678426
- [Background] Sjonnesen K, Berzins S, Fiest KM, M Bulloch AG, Metz LM, Thombs BD, Patten SB. Evaluation of the 9-item Patient Health Questionnaire (PHQ-9) as an assessment instrument for symptoms of depression in patients with multiple sclerosis. Postgrad Med. 2012 Sep;124(5):69-77. doi: 10.3810/pgm.2012.09.2595. PMID 23095427
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Hohol MJ, Orav EJ, Weiner HL. Disease steps in multiple sclerosis: a longitudinal study comparing disease steps and EDSS to evaluate disease progression. Mult Scler. 1999 Oct;5(5):349-54. doi: 10.1177/135245859900500508. PMID 10516779
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] McKay KA, Ernstsson O, Manouchehrinia A, Olsson T, Hillert J. Determinants of quality of life in pediatric- and adult-onset multiple sclerosis. Neurology. 2020 Mar 3;94(9):e932-e941. doi: 10.1212/WNL.0000000000008667. Epub 2019 Nov 15. PMID 31732567
- [Background] Strober LB, Bruce JM, Arnett PA, Alschuler KN, DeLuca J, Chiaravalloti N, Lebkuecher A, Di Benedetto M, Cozart J, Thelen J, Guty E, Roman CAF. Tired of not knowing what that fatigue score means? Normative data of the Modified Fatigue Impact Scale (MFIS). Mult Scler Relat Disord. 2020 Nov;46:102576. doi: 10.1016/j.msard.2020.102576. Epub 2020 Oct 13. PMID 33296974
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Rizzo MA, Hadjimichael OC, Preiningerova J, Vollmer TL. Prevalence and treatment of spasticity reported by multiple sclerosis patients. Mult Scler. 2004 Oct;10(5):589-95. doi: 10.1191/1352458504ms1085oa. PMID 15471378
- [Background] Learmonth YC, Motl RW, Sandroff BM, Pula JH, Cadavid D. Validation of patient determined disease steps (PDDS) scale scores in persons with multiple sclerosis. BMC Neurol. 2013 Apr 25;13:37. doi: 10.1186/1471-2377-13-37. PMID 23617555
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Williams KG, Sanderson M, Jette N, Patten SB. Validity of the Patient Health Questionnaire-9 in neurologic populations. Neurol Clin Pract. 2020 Jun;10(3):190-198. doi: 10.1212/CPJ.0000000000000748. Epub 2020 Apr 13. PMID 32642320
- [Background] Patten SB, Burton JM, Fiest KM, Wiebe S, Bulloch AG, Koch M, Dobson KS, Metz LM, Maxwell CJ, Jette N. Validity of four screening scales for major depression in MS. Mult Scler. 2015 Jul;21(8):1064-71. doi: 10.1177/1352458514559297. Epub 2015 Jan 12. PMID 25583846
- [Background] Olascoaga J. [Quality of life and multiple sclerosis]. Rev Neurol. 2010 Sep 1;51(5):279-88. Spanish. PMID 20669127
- [Background] Rothwell PM, McDowell Z, Wong CK, Dorman PJ. Doctors and patients don't agree: cross sectional study of patients' and doctors' perceptions and assessments of disability in multiple sclerosis. BMJ. 1997 May 31;314(7094):1580-3. doi: 10.1136/bmj.314.7094.1580. PMID 9169401
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Hobart J. Rating scales for neurologists. J Neurol Neurosurg Psychiatry. 2003 Dec;74 Suppl 4(Suppl 4):iv22-iv26. doi: 10.1136/jnnp.74.suppl_4.iv22. No abstract available. PMID 14645463
- [Background] Fayers, P. M. and D. Machin. Quality of life: the assessment, analysis and interpretation of patient-reported outcomes [Internet]. Chichester (England); Hoboken (NJ): John Wiley & Sons, 2007 [cited 2021 June 29]. Available from: https://onlinelibrary.wiley.com/doi/book/10.1002/9780470024522
- [Background] Carroll CA, Fairman KA, Lage MJ. Updated cost-of-care estimates for commercially insured patients with multiple sclerosis: retrospective observational analysis of medical and pharmacy claims data. BMC Health Serv Res. 2014 Jul 2;14:286. doi: 10.1186/1472-6963-14-286. PMID 24986083
- [Background] Coleman CI, Sidovar MF, Roberts MS, Kohn C. Impact of mobility impairment on indirect costs and health-related quality of life in multiple sclerosis. PLoS One. 2013;8(1):e54756. doi: 10.1371/journal.pone.0054756. Epub 2013 Jan 23. PMID 23355896
- [Background] Ney JP, Johnson B, Knabel T, Craft K, Kaufman J. Neurologist ambulatory care, health care utilization, and costs in a large commercial dataset. Neurology. 2016 Jan 26;86(4):367-74. doi: 10.1212/WNL.0000000000002276. Epub 2015 Dec 23. PMID 26701378
- [Background] The Lancet Neurology. Patient-reported outcomes in the spotlight. Lancet Neurol. 2019 Nov;18(11):981. doi: 10.1016/S1474-4422(19)30357-6. No abstract available. PMID 31609205
- [Background] Ponzio M, Gerzeli S, Brichetto G, Bezzini D, Mancardi GL, Zaratin P, Battaglia MA. Economic impact of multiple sclerosis in Italy: focus on rehabilitation costs. Neurol Sci. 2015 Feb;36(2):227-34. doi: 10.1007/s10072-014-1925-z. Epub 2014 Aug 11. PMID 25109816
- [Background] Prescott JD, Factor S, Pill M, Levi GW. Descriptive analysis of the direct medical costs of multiple sclerosis in 2004 using administrative claims in a large nationwide database. J Manag Care Pharm. 2007 Jan-Feb;13(1):44-52. doi: 10.18553/jmcp.2007.13.1.44. PMID 17269836
- [Background] Borreani C, Bianchi E, Pietrolongo E, Rossi I, Cilia S, Giuntoli M, Giordano A, Confalonieri P, Lugaresi A, Patti F, Grasso MG, de Carvalho LL, Palmisano L, Zaratin P, Battaglia MA, Solari A; PeNSAMI project. Unmet needs of people with severe multiple sclerosis and their carers: qualitative findings for a home-based intervention. PLoS One. 2014 Oct 6;9(10):e109679. doi: 10.1371/journal.pone.0109679. eCollection 2014. PMID 25286321
- [Background] Buchanan RJ, Huang C. Informal caregivers assisting people with multiple sclerosis: factors associated with the strength of the caregiver/care recipient relationship. Int J MS Care. 2011 Winter;13(4):177-87. doi: 10.7224/1537-2073-13.4.177. PMID 24453723
- [Background] Holland NJ, Schneider DM, Rapp R, Kalb RC. Meeting the needs of people with primary progressive multiple sclerosis, their families, and the health-care community. Int J MS Care. 2011 Summer;13(2):65-74. doi: 10.7224/1537-2073-13.2.65. PMID 24453707
- [Background] Le Fort M, Wiertlewski S, Bernard I, Bernier C, Bonnemain B, Moreau C, Nicolas-Chouet C, Pavillon T, Tanguy E, Villard A, Bertout P, Bodic P, Desjobert S, Kieny P, Lejeune P, Lombrail P; RESEP-Loire. Multiple sclerosis and access to healthcare in the Pays de la Loire region: preliminary study based on 130 self-applied double questionnaires. Ann Phys Rehabil Med. 2011 May;54(3):156-71. doi: 10.1016/j.rehab.2011.02.005. Epub 2011 Apr 6. English, French. PMID 21515103
- [Background] Lorefice L, Mura G, Coni G, Fenu G, Sardu C, Frau J, Coghe G, Melis M, Marrosu MG, Cocco E. What do multiple sclerosis patients and their caregivers perceive as unmet needs? BMC Neurol. 2013 Nov 15;13:177. doi: 10.1186/1471-2377-13-177. PMID 24237586
- [Background] Matti AI, McCarl H, Klaer P, Keane MC, Chen CS. Multiple sclerosis: patients' information sources and needs on disease symptoms and management. Patient Prefer Adherence. 2010 Jun 24;4:157-61. doi: 10.2147/ppa.s10824. PMID 20622916
- [Background] Mehr SR, Zimmerman MP. Reviewing the Unmet Needs of Patients with Multiple Sclerosis. Am Health Drug Benefits. 2015 Nov;8(8):426-31. PMID 26702334
- [Background] Ponzio M, Tacchino A, Zaratin P, Vaccaro C, Battaglia MA. Unmet care needs of people with a neurological chronic disease: a cross-sectional study in Italy on Multiple Sclerosis. Eur J Public Health. 2015 Oct;25(5):775-80. doi: 10.1093/eurpub/ckv065. Epub 2015 Mar 30. PMID 25829501
- [Background] Solaro C, Ponzio M, Moran E, Tanganelli P, Pizio R, Ribizzi G, Venturi S, Mancardi GL, Battaglia MA. The changing face of multiple sclerosis: Prevalence and incidence in an aging population. Mult Scler. 2015 Sep;21(10):1244-50. doi: 10.1177/1352458514561904. Epub 2015 Jan 12. PMID 25583850
- [Background] Strupp J, Romotzky V, Galushko M, Golla H, Voltz R. Palliative care for severely affected patients with multiple sclerosis: when and why? Results of a Delphi survey of health care professionals. J Palliat Med. 2014 Oct;17(10):1128-36. doi: 10.1089/jpm.2013.0667. Epub 2014 Jul 28. PMID 25068391
- [Background] Young L, Healey K, Charlton M, Schmid K, Zabad R, Wester R. A home-based comprehensive care model in patients with Multiple Sclerosis: A study pre-protocol. F1000Res. 2015 Sep 18;4:872. doi: 10.12688/f1000research.7040.1. eCollection 2015. PMID 26673815
- [Background] Wynia K, Annema C, Nissen H, De Keyser J, Middel B. Design of a Randomised Controlled Trial (RCT) on the effectiveness of a Dutch patient advocacy case management intervention among severely disabled Multiple Sclerosis patients. BMC Health Serv Res. 2010 May 27;10:142. doi: 10.1186/1472-6963-10-142. PMID 20507600
- [Derived] Chu NY, Jamali A, Al Hamarneh YN, Watson KE, Tsuyuki RT, Smyth PS. Provider Experiences With Systematically Administered Patient-Reported Outcome Measures in Multiple Sclerosis: A Qualitative Sub-Study. Neurol Clin Pract. 2025 Aug;15(4):e200486. doi: 10.1212/CPJ.0000000000200486. Epub 2025 Jul 11. PMID 40656127
- [Derived] Chu NY, Yushko L, Pan B, Hamarneh YNA, Watson KE, Tsuyuki RT, Smyth P. Evaluating the impact of systematic reporting of patient-reported outcome measures on depression and anxiety levels in people with multiple sclerosis: a randomized controlled trial. Mult Scler Relat Disord. 2025 Jul;99:106502. doi: 10.1016/j.msard.2025.106502. Epub 2025 May 4. PMID 40339265
- [Derived] Chu NY, Watson KE, Al Hamarneh YN, Yushko L, Tsuyuki RT, Smyth P. Evaluating the impact of patient-reported outcome measures on depression and anxiety levels in people with multiple sclerosis: a study protocol for a randomized controlled trial. BMC Neurol. 2023 Feb 2;23(1):53. doi: 10.1186/s12883-023-03090-0. PMID 36732694
- See also: Atlas of MS 2013: mapping MS around the world (2013) Retrieved June 20, 2021 — https://www.msif.org/wp-content/uploads/2014/09/Atlas-of-MS.pdf
- See also: The way forward: Alberta's multiple sclerosis partnership (2013). Retrieved June 30, 2021 — http://open.alberta.ca/publications/9781460108574